CLINICAL TRIAL: NCT00771979
Title: A Phase I, Randomised, Open-Label, Cross-Over, Single Centre Study in Healthy Volunteers to Determine the Relative Bioavailability of the Phase III Tablet Formulation to the Phase II Tablet Formulation of AZD0530
Brief Title: Relative Bioavailability of Phase II and Phase III Formulations of AZD0530
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mary Stuart, MD, Medical Science Director, Emerging Product Team 1, Oncology, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D8180C00033
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: Healthy Volunteers; Relative Bioavailability
MeSH Terms: interventions — saracatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AZD0530

INTERVENTIONS:
Drug: AZD0530 — of both the Phase II and Phase III AZD0530 125mg tablet variants (A and B) in a random order.
Drug: AZD0530 — Part II: Single doses of AZD0530 125mg oral solution and 2 out of 4 125mg tablet variants (C, D, E and F) in a random order.

SUMMARY:
The aim of the study is to compare how different formulations of AZD0530 are absorbed by the body. As for all clinical trials, safety and tolerability of the drug will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects must be of Non- child-bearing potential
* Body mass index between 19 and 30 kg/m2 and weigh between 50-100 kg

Exclusion Criteria:

* Presence of any clinically significant illness
* Abnormal vital signs
* History of any conditions that may put the subject at risk by participating in the study
* Participation in another clinical study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-11; Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To compare the pharmacokinetic parameters for AZD0530 when administered as Phase III formulation in relation to Phase II formulation. | Pre-dose sample, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72, 120, 168 hours post dose samples.

SECONDARY OUTCOMES:
To monitor the safety of all subjects by assessment of vital signs, ECG, clinical chemistry, haematology, urinalysis and adverse events. | From time of consent to last visit.
An exploratory objective is to characterise the Pharmacokinetic profile of an oral solution of AZD0530 and 4 additional tablet variants of the Phase III formulation of AZD0530 | Pre-dose sample, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72, 120, 168 hours post dose samples.

CONTACTS AND LOCATIONS:
Overall Officials: Raj Chetty, MD, Principal Investigator — AstraZeneca, Clinical Pharmacology Unit, Alderley Park; Mary Stuart, MD, Study Director — AstraZeneca,Parklands, Alderley Park
Locations (1):
- Research Site, Alderley Park, United Kingdom